CLINICAL TRIAL: NCT05007210
Title: The Effects of the One Hour-Whole Body Prenatal Massage Therapy Session on Prenatal Distress and Prenatal Attachment for Women and Their Fetuses During Late Pregnancy: A Randomized Controlled Experimental Trial
Brief Title: The Effects of Whole Body Prenatal Massage Therapy During Pregnancy: A Randomized Controlled Experimental Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Yeliz CAKIR KOCAK, Midwifery Research Asistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Yeliz Çakır Koçak; 16-ASYO-017 (Other Grant/Funding Number: EGE UNIVERSITY)
Record Dates: First submitted 2021-05-18; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Massage Therapy; Pregnancy Related; Fetus Fetus
Keywords: Prenatal massage therapy; Pregnant woman; Fetus; Massage Therapy; Prenatal Distress; Prenatal Attachment; Midwife; Nurse
MeSH Terms: conditions — Fetus-in-Fetu

STUDY DESIGN:
Intervention Model Description: The study type is interventional.As a prospective, randomised, single masking, parallel trial design has been carried out with primipar pregnant women that came to obstetrics polyclinic of a university hospital to evaluate before 30th week.The participants were randomly allocated to the parallel comparison groups by a central office.The sample selection process in the study has been applied according to CONSORT criteria (Moher et al. 2010), and through the permutation method, blocked randomization (Kanık, Tasdelen, and Erdogan 2011) has been done to the records assigned from the centre that the study was applied. The completion decision of the data gathering process has been determined with power analysis that is carried out by the PASS program.
Who Masked: Outcomes Assessor
Masking Description: The pregnant women in control and prenatal massage therapy groups were appointed to different times to avoid each other. At the beginning of the study, they didn't know in which group they were taken to participate in the study. In the process of gathering data, the single-blind method has been applied, and the double-blind method has only been applied to data analysis (The double-blind method was not used in the data collection process in order to reveal the loss of the study conducted within the scope of the doctoral thesis and the fact that prenatal massage therapy practice is not performed routinely in country conditions). However, single blinding was performed in terms of the outcomes. The data obtained from the research were analyzed by Biostatistics and Medical Information Department at Ege University.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal massage therapy group (Experimental): Prenatal massage therapy for prenatal attachment, physiological and psychological distress, maternal and fetal well-being.
  Interventions: Other: Prenatal massage therapy
- Control group (No Intervention): Pregnant women in the control group were interviewed twice (once a week for 30th and 34th week) by the same massaging midwife. No additional attempt was made except for filling out the forms and evaluating the biophysical profile by the obstetrician in these interviews. The massaging midwife's phone number was given to the pregnant women in both groups if they want to reach anytime. A phone number was set for the study, and this phone number was used by the massaging midwife. This service has been provided for pregnant women to reach her whenever they want.

INTERVENTIONS:
Other: Prenatal massage therapy — Pregnant women in the intervention group had a whole body prenatal massage therapy every week between 30th and 34th gestational weeks (once a week, 5-weeks in total and 60-minutes each).Session content for the prenatal massage therapy group was created by the researcher who was 640-hours trained massaging midwife.It included 12 different massage techniques (Osborne 2015, Osborne 2021).Also, the session, which included deep tissue and Sweden massage methods, had been applied.Each session began with the pregnant woman in a side-lying position with standart special pillows (30-minutes for left, 30-minutes for right).EFM, BPP, vital signs, FHR evaluation were carried out for all participants per visiting the hospital for the study.BPP before and after prenatal massage therapy was evaluated by an obstetrician.A phone number was set for the study, and this phone number was used by the massaging midwife.The service has been provided for pregnant women to reach her whenever they want.
  Arms: Prenatal massage therapy group

SUMMARY:
Background: Massage therapy in many parts of the world is used in all periods of pregnancy.

Aim: The study aimed to determine the effect of massage therapy during pregnancy on women and their fetuses in a university hospital in Izmir, Turkey.

Method: A randomized controlled experimental trial was aimed to reach primipara pregnant women, 20-35 years old, who came to a university obstetric clinic to get the results of the first-trimester screen test. Researchers aimed to reach 30 pregnant women at the start of the study. Participants were randomly allocated to a parallel comparison group by a central office. The sampling technique has been applied according to the CONSORT criteria.

The study practices have been carried out after receiving ethics committee and institution approvals after the researcher completed the prenatal massage therapy training, and after taking the voluntary informed consent of the pregnant women. The practices have been carried out in the massage office that was formed within the scope of the study. Electronic fetal monitoring (EFM), BPP, vital signs, fetal heart rate (FHR) evaluation have been carried out for the pregnants whose routine gestational monitoring went on during their gestational week between the 30th and 34th in the control group, and Pregnant Description Form, VAS, Prenatal Attachment Inventory-PAI, Revised Prenatal Distress Questionnaire-PDQ have been applied. In the prenatal massage therapy group, between the 30th and 34th weeks, each week for five weeks, prenatal massage therapy including a 60 minutes deep tissue and Sweden massage methods had been applied once a week. Side-Lying Positioning System that is designed specifically for the pregnant has been used during the practices. In addition, the reason why the study group consisted of pregnant women in these weeks; Perinatology specialists recommend women to experience a deep and sustainable level of relaxation for 45-60 minutes before falling asleep, especially in the last 6-8 weeks of pregnancy, in preparation for labour (Osborne et al. 2021). In line with this suggestion, since the whole body massage has been performed in the research method, a 60-minute massage (30 minutes for each lateral position) has been applied.

DETAILED DESCRIPTION:
Aim: The study aims to determine the effect of massage during pregnancy on women and their fetuses in a university hospital in Izmir, Turkey.

Method: The study was a randomized controlled experimental trial carried out with 20-35 years-old primipara pregnant women who came to obstetrics polyclinic of a university for evaluation of their first-trimester screen test's results, had no infertility story and were not at high risk (inclusion criteria). The participants were randomly allocated to the parallel comparison groups by a central office. The sample selection process in the study has been planned to be applied according to the CONSORT criteria (Moher et al. 2010) and the permutation method with blocked randomization has been done to the records assigned from the centre that the study was applied (Kanık, Tasdelen, and Erdogan 2011). In the process of collecting data, one blinding method has been applied, and it has only been applied to data analysis. Researchers aimed to reach 30 pregnant women at the start of the study. The completion decision of the data gathering process has been determined with power analysis that is carried out by the PASS program.

The study practices have been carried out after receiving ethics committee and institution approvals after the researcher completed the prenatal massage therapy training, and after taking the voluntary informed consent of the pregnant women. The practices have been carried out in the massage office that was formed within the scope of the study. Electronic fetal monitoring (EFM), BPP, vital signs, fetal heart rate (FHR) evaluation have been carried out for the pregnants whose routine gestational monitoring went on during their gestational week between the 30th and 34th in the control group, and Pregnant Description Form, VAS, Prenatal Attachment Inventory-PAI, Revised Prenatal Distress Questionnaire-PDQ have been applied. In the prenatal massage therapy group, between the 30th and 34th weeks, each week for five weeks, prenatal massage therapy including a 60 minutes deep tissue and Sweden massage methods had been applied once a week. Side-Lying Positioning System that is designed specifically for the pregnant has been used during the practices. In addition, the reason why the study group consisted of pregnant women in these weeks; Perinatology specialists recommend women to experience a deep and sustainable level of relaxation for 45-60 minutes before falling asleep, especially in the last 6-8 weeks of pregnancy, in preparation for labour (Osborne et al. 2021). In line with this suggestion, since the whole body massage has been performed in the research method, a 60-minute massage (30 minutes for each lateral position) has been applied.

Like before the prenatal massage therapy on the first date and after the prenatal massage therapy on the last date in the control group, all the forms and measurements have been applied. Pregnant women's VAS was measured before and after the prenatal massage therapy and the evaluation of the other measured data have been held between the 31st and 33rd gestational weeks. Also, Visual Analog Patient Satisfaction Scale-VAPSS has been measured after each prenatal massage therapy for finding satisfaction levels. In the process of the study, any significant side effect related to the practices hasn't occurred. The completion decision of the data gathering process has been determined with power analysis that was carried out by PASS program. The analysis of the study data has been carried out through SPSS 16 program.

ELIGIBILITY:
Inclusion Criteria:

* 20-35 years-old
* Primiparous women
* Low-risk pregnant women
* Before the 30th week of gestation Also for the group of the prenatal massage therapy;
* Can come 5 times for each week of gestation between 30 and 34 weeks
* No infectious disease or skin infection on the skin,
* No thrombosis or phlebitis
* Single and healthy fetus
* Written and verbally available
* Before the 30th week of gestation
* Accept attendance
* Residing in the province in which the study conducted city

Exclusion Criteria:

* Infertility story
* High risk pregnancy
* Live or stillbirth after 20th week of gestation
* Abortion after the first trimester
* History of recurrent pregnancy loss

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Prenatal Attachment Inventory (PAI): | from 30 weeks up to 34 weeks
  The scale was developed by Muller (1993) and its Turkish validity-reliability study was carried out by Dereli Yılmaz and Kızılkaya Beji (2013). It is used to explain women's thoughts, feelings and situations during pregnancy and to determine the level of attachment to the baby in the prenatal period. Increased score from the scale shows that the prenatal attachment level increases. Cronbach alpha reliability coefficients ranged from 0.81 (Muller 1993) and 0.84 (Dereli Yilmaz and Kızılkaya Beji 2013). The internal reliability of this instrument was 0.87 for 30th week and 0.90 for 34th week in this sample.
Revised Prenatal Distress Questionnaire (NuPDQ): | from 30 weeks up to 34 weeks
  The scale with different versions was developed by Yali and Lobel and the version of 17-item NuPDQ was revised by Lobel et al. (Lobel 2008; Yali and Lobel 1999). Its Turkish validity-reliability study was carried out by Yüksel et all. (Yüksel, Akın, and Durna 2011). It evaluates difficulties in pregnancy which about specific concerns and anxieties specific to the pregnancy period, such as medical problems, physical symptoms, parenting, relationships, bodily changes, birth and baby's health. The reduction of the total score of the scale shows that the prenatal distress level perceived by pregnant women decreases. Cronbach alpha reliability coefficients ranged from 0.79-0.88 (Ibrahim and Lobel 2020) and 0.85 (Yüksel et al. 2011). The internal reliability of this instrument was 0.73 for 30th week and 0.85 for 34th week in this sample.

SECONDARY OUTCOMES:
Maternal hearth rate (MHR): | from 30 weeks up to 34 weeks
  It was carried out for all pregnant women (control and prenatal massage therapy groups) per visiting the hospital for the study by the same midwife. The assessment were made before and after the prenatal massage therapy sessions on the first and last days of the 5-week study (two times for the control group and 10 times for the prenatal massage therapy group between the 30th and 34th gestational weeks).
Fetal hearth rate (FHR): | from 30 weeks up to 34 weeks
  It was carried out for all pregnant women (control and prenatal massage therapy groups) per visiting the hospital for the study by the same midwife. The assessment were made before and after the prenatal massage therapy sessions on the first and last days of the 5-week study (two times for the control group and 10 times for the prenatal massage therapy group between the 30th and 34th gestational weeks).
Biophysical Profile (BPP): | from 30 weeks up to 34 weeks
  BPP is a prenatal test used to measure the health of fetus. It has a procedure in which some variables in the USG (fetal breathing movement, fetal body movement, fetal muscle tone, amniotic fluid volume, fetal heart rate reaction) is assessed. The highest score that can be obtained from the BFP assessment is 10 (≤4: abnormal, 6: doubtful, 8-10: normal) (Alp Dal and Ertem 2016). It was carried out for all pregnant women (control and prenatal massage therapy groups) per visiting the hospital for the study by the same obstetrician. The assessment were made before and after the prenatal massage therapy sessions on the first and last days of the 5-week study (two times for the control group and 10 times for the prenatal massage therapy group between the 30th and 34th gestational weeks).
Visual Analog Scale (VAS): | from 30 weeks up to 34 weeks
  It is developed and high reliability have been found by Hayes and Patterson. Its advantages are quickly filled out, simple, interesting, easily scored, the rater is freed from quantitative terms, it requires no master scale (Hayes and Patterson 1921). It is used to make some values that do not measure numerically. The scale is used in many different areas of health. Its main advantage is that it does not have a language and is easy to apply and consisting of a single 100 mm line (Clarke 1964). Cline et al. (1992) found that the vertical use of it is better understood (Cline et al. 1992). The mean value obtained for individuals in the general assessment is taken. Turkish validity and reliability study conducted by Eti Aslan and it is quite reliable in literate group (Eti Aslan 2004). Evaluation was performed over vertical 100 mm measurement in the study.
Visual Analog Patient Satisfaction Scale-VAPSS: | from 30 weeks up to 34 weeks
  Kılınçer ve Zileli (2006) combined two scales features (Visual Analog Pain Scale and Wong-Baker Scale) and arranged VAPSS. It is a measurement tool that can be applied for individuals and all ages also all culture levels. They reported that the scale can use in pregnant women (Kılınçer and Zileli 2006). Evaluation was performed over vertical 100 mm measurement in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeliz Çakır Koçak, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alp Dal, N., & Ertem, G. (2016). Fetal Sağlığın Değerlendirilmesi ve Tarama Testleri. In Ü. Sevil & G. Ertem (Eds.), Perinatoloji ve Bakım (Birinci ba, pp. 373-408). Ankara Nobel Tıp Kitabevleri.
- [Background] Clarke, M. (1964). Reliability and sensibility in the self-assessment of well-being. Bul Br Psy Soc, 17(18A).
- [Background] Cline ME, Herman J, Shaw ER, Morton RD. Standardization of the visual analogue scale. Nurs Res. 1992 Nov-Dec;41(6):378-80. No abstract available. PMID 1437591
- [Background] Dereli Yilmaz, S., & Kızılkaya Beji, N. (2013). Prenatal Bağlanma Envanterinin Türkçe'ye Uyarlanması: Güvenilirlik ve Geçerlilik Çalışması. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 16(2), 103-109.
- [Background] Eti Aslan, F. (2004). Ameliyat Sonrası Ağrı Değerlendirmesinde Görsel Kıyaslama Ölçeğiyle Basit Tanımlayıcı Ölçeğin Duyarlık ve Seçiciliği. Yoğun Bakım Hemşireliği Dergisi, 8(1), 1-6. http://dergipark.gov.tr/ybhd/issue/26499/278822
- [Background] Hayes, M. H. S., & Patterson, D. G. (1921). Experimental development of the graphic rating method. Psychological Bulletin, 18, 98-99.
- [Background] Ibrahim SM, Lobel M. Conceptualization, measurement, and effects of pregnancy-specific stress: review of research using the original and revised Prenatal Distress Questionnaire. J Behav Med. 2020 Feb;43(1):16-33. doi: 10.1007/s10865-019-00068-7. Epub 2019 Jun 10. PMID 31183596
- [Background] Kanık, E. A., Tasdelen, B., & Erdogan, S. (2011). Randomization In Clinical Trials. Marmara Medical Journal, 24, 149-155. https://doi.org/10.5472/MMJ.2011.01981.1
- [Background] Kılınçer, C., & Zileli, M. (2006). Görsel Analog Hasta Tatmini Skalası. Trakya Univ Tip Fak Derg, 23(3), 113-118.
- [Background] Lobel M, Cannella DL, Graham JE, DeVincent C, Schneider J, Meyer BA. Pregnancy-specific stress, prenatal health behaviors, and birth outcomes. Health Psychol. 2008 Sep;27(5):604-15. doi: 10.1037/a0013242. PMID 18823187
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Muller ME. Development of the Prenatal Attachment Inventory. West J Nurs Res. 1993 Apr;15(2):199-211; discussion 211-5. doi: 10.1177/019394599301500205. No abstract available. PMID 8470375
- [Background] Osborne, C. (2015). Pre- and Perinatal Massage Therapy Certification Workshop Student Guide (Special Document).
- [Background] Yali AM, Lobel M. Coping and distress in pregnancy: an investigation of medically high risk women. J Psychosom Obstet Gynaecol. 1999 Mar;20(1):39-52. doi: 10.3109/01674829909075575. PMID 10212886
- [Background] Yüksel, F., Akın, S., & Durna, Z. (2011). "Prenatal Distres Ölçeği"nin Türkçe'ye Uyarlanması ve Faktör Analizi. Hemşirelikte Eğitim ve Araştırma Dergisi, 8(3), 43-51.
- [Result] Osborne, C., Kolakowski, M., & Lobenstine, D. M. (2021). Pre- and Perinatal Massage Therapy (M. Law & W. Lee (eds.); Third edit). Handspring Publishing Limited. https://www.handspringpublishing.com/product/pre-and-perinatal-massage-third-edition/